CLINICAL TRIAL: NCT01449890
Title: Randomized Trial of E-mail Follow-up Care After Cognitive Behavioural Treatment for Depression
Brief Title: Randomized Trial of Depression Follow-up Care by Email
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, PD Dr. phil. Birgit Watzke, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRV0422/00-40-65-50-24
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Depressive Disorders
Keywords: follow up care; e-mail; effectiveness; depressive disorders
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- E-mail follow up care (Experimental): After having terminated inpatient CBT patients receive follow up care by email for 12 weeks (on average one contact per week). The follow up care aims at supporting the patients in continuing exercises they have learned during the initial treatment phase in order to cope with depression, e.g. integrating positive activities in their all day life or monitoring the interdependence of cognition, emotion and behaviour.
  Interventions: Behavioral: E-mail follow up care
- Treatment as usual (No Intervention): After having terminated inpatient CBT patients receive treatment as usual within routine care.

INTERVENTIONS:
Behavioral: E-mail follow up care — After having terminated inpatient CBT patients receive follow up care by email for 12 weeks (on average one contact per week). The follow up care aims at supporting the patients in continuing exercises in order to cope with depression.
  Other Names: internet based psychotherapy; web based psychotherapy
  Arms: E-mail follow up care

SUMMARY:
The primary objective of this study is to test in a randomized effectiveness trial if e-mail delivered cognitive behavioural treatment is an effective follow-up care approach in the treatment of depression under clinically representative conditions.

DETAILED DESCRIPTION:
Depression belongs to the most prevalent mental disorders and often goes along with a high burden of disease. Although the efficacy and the effectiveness of psychological treatments for depressive disorders have been demonstrated, there remains the problem of maintaining the benefits achieved during the initial treatment phase. Therefore options of follow-up care have to be considered. Since access to psychotherapeutic treatments is limited and costly, internet-based interventions can offer a feasible opportunity for follow-up care in order to enhance the long-term effectiveness of psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Depressive disorder: F32.0-F32.2; F33.0-F33.2; F34.1 according to ICD-10
* Precursory CBT
* Internet access

Exclusion Criteria:

* No knowledge of the German language
* Risk of suicide
* Acute psychosis or psychotic symptoms
* Established concurrent in vivo CBT after discharge from inpatient CBT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Measure of the severity of depression - Beck Depression Inventory (BDI- II) | Change in the BDI-II from baseline (beginning of treatment) to follow up (3 months after termination of the follow-up care)

SECONDARY OUTCOMES:
Measure of health related quality of life - SF-8 | Change in the SF-8 from baseline (beginning of treatment) to follow up (3 months after termination of the follow-up care
  SF-8: short version of the SF -36
GAD-7 | Change in the GAD-7 from baseline (beginning of treatment) to follow up (3 months after termination of the follow-up care)
  Measure for generalized anxiety disorder
Depressive relapse/recurrence | Measured at follow up (3 months after termination of the follow-up care)

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Watzke, PhD, Principal Investigator — University Medical Center Hamburg-Eppendorf Centre of Psychosocial Medicine Department of Medical Psychology
Locations (1):
- University Medical Center Hamburg-Eppendorf, Centre of Psychosocial Medicine, Department of Medical Psychology, Hamburg, Hamburg, Germany